CLINICAL TRIAL: NCT02749357
Title: Effect of Different Programs of Robotic Assisted Gait Training in Individuals With Chronic Motor Incomplete Spinal Cord Injury.
Brief Title: Robotic Gait Training in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Jimena Quinzaños, Chief of Neurologic Rehabilitation Department, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35/15
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injuries
Keywords: gait; robotic orthosis
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Intervention: Control group, with 30 training sessions in robotic orthosis with duration of 30 minutes during 6 weeks.
  The initial training speed will be the comfortable one for each patient, as assessed by Swinnen.The training progression will consist in a 10% weekly increase in speed, and a 5% weekly reduction of partial weight support.
  Interventions: Device: 30 minutes Lokomat
- Experimental (Experimental): Intervention: Experimental group, with 30 training sessions in robotic orthosis with duration of 60 minutes during 6 weeks.
  The initial training speed will be the comfortable one for each patient, as assessed by Swinnen.The training progression will consist in a 10% weekly increase in speed, and a 5% weekly reduction of partial weight support.
  Interventions: Device: 60 minutes Lokomat

INTERVENTIONS:
Device: 30 minutes Lokomat — 30 training sessions in robotic orthosis with duration of 30 or 60 minutes during 6 weeks, duration of 30 minutes.
  The initial training speed will be the comfortable one for each patient, as assessed by Swinnen (20). The training progression will consist in a 10% weekly increase in speed, and a 5% weekly reduction of partial weight support.
  Arms: Control
Device: 60 minutes Lokomat — 30 training sessions in robotic orthosis with duration of 30 or 60 minutes during 6 weeks, duration of 60 minutes.
  Arms: Experimental

SUMMARY:
INTRODUCTION:

The ability to move and transfer own body in an effective manner, is frequently affected in people with a spinal cord injury with a negative impact in mood and quality of life, in such a way, that achieving an effective locomotion, is one of the main objectives in the rehabilitation program in a spinal cord injured patient.

There are different modalities of locomotion training in spinal cord injury, being the robotic orthosis among them, and offering until now, positive outcomes. However there´s still a lack of evidence of the optimal training characteristics, in order to establish the best time, number of sessions, and progression scheme. For these reasons, establishing the effects of different locomotion training programs will provide the necessary data in order to develop an effective training program for the maximum benefit of the patient.

OBJECTIVE To determine the effect of different training programs with robotic gait orthosis for patients with chronic motor incomplete spinal cord injury (SCI) (American Spinal Injury Association Impairment Scale (AIS) C / D) in short and long term.

METHODS AND DESIGN. The design of the study consists on a randomized, blinded to the observer, clinical trial.

Patients from the National Institute of Rehabilitation (INR) with spinal cord injury, AIS C and D, with at least 6 months of evolution, and who are able to walk with or without gait auxiliary, will be eligible.

Informed consent will be obtained from all subjects prior to participation. Patients will be randomly assigned to either one of the two different training groups: intervention or control group.

The control group will be submitted to training sessions of 30 minutes, and the intervention group will have training sessions of 60 minutes.

Both groups will receive a training period of six weeks, five days a week.

Throughout the training period, gait assessments with the GaitRite instrument, will be performed, and repeated at 6 and 12 months after completion of the training as part of follow up. The data obtained from the GaitRite will be compared within each group, in order to determine which type of training is more effective

Statistical analysis will be performed using SPSS, considering all P < 0.05 as statistically significant.

DETAILED DESCRIPTION:
A Spinal cord injury (SCI) is the disruption of the nerve pathways that connect the brain to the rest of the body, causing the cessation of their motor, sensory and vegetative functions. It is considered one of the most devastating clinical conditions affecting the functionality and independence of the individual.

The World Health Organization estimates an annual overall incidence of 40-80 new cases per million, equivalent to 250 000 to 500 000 individuals with spinal cord injury each year. The consequences of the SCI, significantly impair the ability of the patient to perform daily life activities, and their overall quality of life.Decreased mobility is the main element that affects lower satisfaction and quality of life. The improvement of mobility or the ability to move in an energy efficient manner improves the quality of life in patients with SCI.

The recovery of walking function is considered of great relevance both by patients and physicians. The most relevant prognostic factor for functional recovery in SCI patients is the neurological status at the moment of the first examination, considering the neurological level and the severity of the lesion according to the American Spinal Injury Association impairment scale (AIS).

According to Scivoletto, of the patients with American Spinal Injury Association (ASIA) impairment scale A, with thoracic and lumbar lesion only 6.4% achieve functional walking. In patients with ASIA B, have an overall rate of ambulation of 23.5%, ASIA C have 51.4% and ASIA D patients have a prognosis for walking recovery between 80-100% (88.9%).

In another study, Dobkin[8] reported that 35% of individuals classified as AIS B, 92% of subjects AIS C and all subjects AIS D recovered the ability to walk after gait training intervention with partial weight bearing for a period of 8 weeks. However, of all the patients with spinal cord injury, few regain a functional gait capacity, due to a low speed, a decreased step length, cadence and changes in rhythm and coordination.

In fact, spinal cord injury often leads to changes in walking patterns, which are associated with postural changes related to poor ability to transfer bodyweight, alterations in balance and equilibrium. Other important factors in the process of walking recovery include: lack of coordination and development of propulsion, sensory loss, and hyperactive spinal reflexes. These deficiencies are severe enough to delay standing and gait rehabilitation process .

Some of the most important gait abnormalities in individuals who suffer spinal cord injuries are: the inability to stand without assistance, the voluntary movement of joints such as hip hip, knee and ankle, knee hyperextension, inability to move the legs without making compensation mechanisms, foot dragging, changes in weight transfer during walking, lack of coordination, transition among phases of gait, and falls.

That is the reason why many gait training programs have been evaluated. Current modalities of gait training, pretend to activate the locomotor center of the central pattern generator by repetitive gait stimuli, allowing the central nervous system plasticity to create new neural pathways and connections in the spinal cord, making possible walking recovery in patients with spinal cord injury. Evidence favors two gait training modalities: the treadmill with partial weight-support and the robotic-assisted gait. These training modalities provide an improvement in gait parameters and functionality when compared to conventional physiotherapy, as shown in the systematic review by Morawietz and Moffat in which different programs of gait training in patients with SCI AIS C and D of diverse etiology of chronic and acute evolution and any neurological level are compared.

Although the use of treadmill , partial weight-bearing and robotic orthotics are essential in the training of locomotion in SCI patients , little has been published about the progress of the training, clinical decision making and evaluation of progress.[16] Most of the studies on the subject provide only very general criteria to optimize treatment (modifying body weight support and speed training), providing insufficient evidence to guide the training progression in parameters such as training frequency, speed and optimal duration of treatment.

As a result, it is important to develop studies which test training strategies that help to clarify issues related to the amount, intensity, frequency, and progression of training in order to achieve the maximum recovery of gait for individuals with SCI. Accordingly, to determine and compare the effect of different gait training programs will orient the development of more effective training programs.

OBJECTIVE

To determine the effects on gait of different gait training programs using a robotic gait orthosis in individuals with chronic incomplete SCI (AIS C/D).

Specific Objectives

1. To evaluate changes in functionality of gait and spatiotemporal gait parameters, functional independence, lower limbs muscle force, spasticity and joint range of motion of individuals according to different progression programs.
2. To determine in the short term (immediately posterior to training program), medium term (6 months) and long term (1 year) effect on individuals' functionality of gait, spatiotemporal gait parameters and functional independence obtained with different gait training programs.
3. To compare the effect of the two different programs of gait training using a robotic gait orthosis.

METHODS

7.1.- Study Design: Randomized Clinical Trial blinded to observer.

7.2.- Subjects: Subjects from inpatient and outpatient services within the Neurologic Rehabilitation Department of the National Institute of Rehabilitation with SCI AIS C and D, with at least 6 months since injury and able to walk with or without walking aids.

Sample Size

Sample Size was calculated based on improvement on gait velocity reported by previous published studies using the program Epidat 4.

It was calculated that 23 patients are required in order to detect a difference between means of 32.3 cm/s, as reported by Wirz , with a standard deviation of 37.5 cm/s, a power of 80% and a confidence level of 95% On the other hand, Hornby reported a difference between means of 0.36 m/s with a standard deviation of 0.14 m/s, which results on a sample size of 4 subjects per group.

Due these differences, an initial trail will performed with an initial sample size of 4 subjects per group and a new calculation of power of the study will be made in order to determine convenience of sample size or necessity of a bigger sample.

RANDOMIZATION The randomization will be conducted by a digital randomization system with atmospheric noise, available at random.org. Allocation will be done by a person not included in the protocol.

Proceeding

The outpatients that assist to the Spinal Cord Injury Service at the "Instituto Nacional de Rehabilitación" will be randomly assigned to two different groups.. The groups are defined as follow:

A. Control group, with 30 training sessions in robotic orthosis with duration of 30 minutes during 6 weeks.

B. Control group, with 30 training sessions in robotic orthosis with duration of 60 minutes during 6 weeks.

Proposed statistical analysis

Descriptive statistics will be carried out with measures of central tendency for quantitative variables and proportions for qualitative variables. In order to analyze differences between groups, co variance analysis will be conducted. We will consider results as statistically significative when p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete SCI AIS C or D with at least 6 months of evolution.
* Any etiology
* Able to walk with or without walking aids.
* Properly signed written informed consent.

Exclusion Criteria:

* Orthopedic conditions like bone instability , arthrodesis
* Metabolic pathology which impedes exercise.
* Audio or visual alterations.
* Own Robotic Orthoses (lokomat) counter-indications: body weight bigger than 135 kg, open lesions in skin of lower extremities or torso, non-cooperative patients, mechanical ventilation or continuum use of oxygen.
* Uncontrolled pain.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05; Primary Completion 2021-06 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Baseline Gait speed | Before training
  Analysed by the Gait Rite system (m/s)
Change in gait speed at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (m/s)
Change in gait speed at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (m/s)
Change in gait speed at third training session | Before and after the third session of training (day3)
  Analysed by the Gait Rite system (m/s)
Change from baseline gait speed at first week | At the end of the first training week
  Analysed by the Gait Rite system (m/s)
Change from baseline gait speed at second week | At the end of the second training week
  Analysed by the Gait Rite system (m/s)
Change from baseline gait speed at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (m/s)
Change from baseline gait speed at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (m/s)
Baseline mean double support percentage | Before training
  Analysed by the Gait Rite system (0-100%)
Change in mean double support percentage at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-100%)
Change in mean double support percentage at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-100%)
Change in mean double support percentage at third training session | Before and after the second session of training (day 3)
  Analysed by the Gait Rite system (0-100%)
Change from baseline mean double support percentage at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline mean double support percentage at second week | At the end of the secondt training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline mean double support percentage at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline mean double support percentage at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline mean double support percentage at six months | At 6 months
  Analysed by the Gait Rite system (0-100%)
Change from baseline mean double support percentage at one year | At one year
  Analysed by the Gait Rite system (0-100%)
Change from baseline gait speed at six months | At 6 months
  Analysed by the Gait Rite system (m/s)
Change from baseline gait speed at one year | At one year
  Analysed by the Gait Rite system (m/s)
Baseline Functional ambulation profile (FAP) | Before training
  Analysed by the Gait Rite system (0-100)
Change in FAP at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-100)
Change in FAP at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-100)
Change in FAP at third training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-100)
Change from baseline FAP at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-100)
Change from baseline FAP at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-100)
Change from baseline FAP at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-100)
Change from baseline FAP at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-100)
Change from baseline FAP at six months | At 6 months
  Analysed by the Gait Rite system (0-100)
Change from baseline FAP at one year | At one year
  Analysed by the Gait Rite system (0-100)
Baseline Mean single support | Before training
  Analysed by Gait Rite System (0-100%)
Change in Mean single support at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-100%)
Change in Mean single support at second training session | Before and after the first session of training (day 2)
  Analysed by the Gait Rite system (0-100%)
Change in Mean single support at third training session | Before and after the first session of training (day 3)
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean single support at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean single support at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean single support at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean single support at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean single support at six months | At 6 months
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean single support at one year | At one year
  Analysed by the Gait Rite system (0-100%)
Baseline Step time | Before training
  Analysed by Gait Rite System (0-10s)
Change in Step time at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-10s)
Change in Step time at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-10s)
Change in Step time at third training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-10s)
Change from baseline Step time at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-10s)
Change from baseline Step time at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-10s)
Change from baseline Step time at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-10s)
Change from baseline Step time at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-10s)
Change from baseline Step time at six months | At 6 months
  Analysed by the Gait Rite system (0-10s)
Change from baseline Step time at one year | At one year
  Analysed by the Gait Rite system (0-10s)
Baseline Step length | Before training
  Analysed by Gait Rite System (0-1m)
Change in Step length at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-1m)
Change in Step length at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-1m)
Change in Step length at first training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step length at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step length at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step length at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system(0-1m)
Change from baseline Step length at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step length at six months | At 6 months
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step length at one year | At one year
  Analysed by the Gait Rite system (0-1m)
Baseline Mean double support | Before training
  Analysed by Gait Rite System (0-100%)
Change in Mean double support at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-100%)
Change in Mean double support at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-100%)
Change in Mean double support at third training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean double support at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean double support at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean double support at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean double support at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean double support at six months | At 6 months
  Analysed by the Gait Rite system (0-100%)
Change from baseline Mean double support at one year | At one year
  Analysed by the Gait Rite system (0-100%)
Baseline Support base width | Before training
  Analysed by Gait Rite System (0-1m)
Change in Support base width at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system(0-1m)
Change in Support base width at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-1m)
Change in Support base width at third training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-1m)
Change from baseline Support base width at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Support base width at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Support base width at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Support base width at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Support base width at six months | At 6 months
  Analysed by the Gait Rite system (0-1m)
Change from baseline Support base width at one year | At one year
  Analysed by the Gait Rite system (0-1m)
Baseline Step width | Before training
  Analysed by Gait Rite System (0-1m)
Change in Step width at first training session | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system(0-1m)
Change in Step width at second training session | Before and after the second session of training (day 2)
  Analysed by the Gait Rite system (0-1m)
Change in Step width at third training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step width at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step width at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step width at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step width at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step width at six months | At 6 months
  Analysed by the Gait Rite system (0-1m)
Change from baseline Step width at one year | At one year
  Analysed by the Gait Rite system (0-1m)
Baseline Variation coefficient of the plantar support´s lenght | Before training
  Analysed by Gait Rite System (0-100%)
Change in Variation coefficient of the plantar support´s lenght at first training sesion | Before and after the first session of training (day 1)
  Analysed by the Gait Rite system (0-100%)
Change in Variation coefficient of the plantar support´s lenght at second training session | Before and after the first session of training (day 2)
  Analysed by the Gait Rite system (0-100%)
Change in Variation coefficient of the plantar support´s lenght at third training session | Before and after the third session of training (day 3)
  Analysed by the Gait Rite system (0-100%)
Change from baseline Variation coefficient of the plantar support´s lenght at first week | At the end of the first training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Variation coefficient of the plantar support´s lenght at second week | At the end of the second training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Variation coefficient of the plantar support´s lenght at fourth week | At the end of the fourth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Variation coefficient of the plantar support´s lenght at the end of the training | At the end of the sixth training week
  Analysed by the Gait Rite system (0-100%)
Change from baseline Variation coefficient of the plantar support´s lenght at six months | At 6 months
  Analysed by the Gait Rite system (0-100%)
Change from baseline Variation coefficient of the plantar support´s lenght at one year | At one year
  Analysed by the Gait Rite system (0-100%)

SECONDARY OUTCOMES:
Baseline Strength | Before training
  Muscular tension necessary to overcome a position or resistance Lokomat L-FORCE (Nm)
Change from baseline Strength at the end of the training | At the end of the sixth training week
  Muscular tension necessary to overcome a position or resistance Lokomat L-FORCE (Nm)
Change from baseline Strength at six months | At 6 months
  Muscular tension necessary to overcome a position or resistance Lokomat L-FORCE (Nm)
Change from baseline Strength at one year | At one year
  Muscular tension necessary to overcome a position or resistance (Nm) Lokomat L-FORCE
Baseline Spasticity | Before training
  Muscular resistance to passive movement related to speed (Nm/°) L-STIFF at 30, 60 and 90°/s
Change from baseline Spasticity at the end of the training | At the end of the sixth training week
  Muscular resistance to passive movement related to speed (Nm/°) L-STIFF at 30, 60 and 90°/s
Change from baseline Spasticity at six months | At 6 months
  Muscular resistance to passive movement related to speed (Nm/°) L-STIFF at 30, 60 and 90°/s
Change from baseline Spasticity at one year | At one year
  Muscular resistance to passive movement related to speed (Nm/°) L-STIFF at 30, 60 and 90°/s
Baseline Range of motion (ROM) | Before training
  Range of motion from an articulation. Lokomat L-ROM (degrees)
Change from baseline Range of motion (ROM) at the end of the training | At the end of the sixth training week
  Range of motion from an articulation. Lokomat L-ROM(degrees)
Change from baseline Range of motion (ROM) at six months | At 6 months
  Range of motion from an articulation. Lokomat L-ROM (degrees)
Change from baseline Range of motion (ROM) at one year | At one year
  Range of motion from an articulation. Lokomat L-ROM (degrees)
Baseline SCIM-III (Spinal Coprd Independence Measure III) | Before training
  Spinal Cord Independence Measure III (Amount of independence in self-care, sphincter control, transference and locomotion activities) (0-100)
Change from baseline SCIM-III at the end of the training | At the end of the sixth training week
  Spinal Cord Independence Measure III (Amount of independence in self-care, sphincter control, transference and locomotion activities) (0-100)
Change from baseline SCIM-III at six months | At 6 months
  Spinal Cord Independence Measure III (Amount of independence in self-care, sphincter control, transference and locomotion activities) (0-100)
Change from baseline SCIM-III at one year | At one year
  Spinal Cord Independence Measure III (Amount of independence in self-care, sphincter control, transference and locomotion activities) (0-100)
Baseline Satisfaction with life | Before training
  Life satisfaction Questionnaire 9 (LISAT 9)(0-36)
Change from baseline Satisfaction with life at the end of the training | At the end of the sixth training week
  Life satisfaction Questionnaire 9 (LISAT 9)(0-36)
Change from baseline Satisfaction with life at six months | At 6 months
  Life satisfaction Questionnaire 9 (LISAT 9)(0-36)
Change from baseline Satisfaction with life at one year | At one year
  Life satisfaction Questionnaire 9 (LISAT 9) (0-36)
Baseline Functioning, Disability and Health classification | Before training
  BRIEF-CORE SET OF THE ICF-CY (International Classification of Functioning, Disability and Health)
Change from baseline Functioning, Disability and Health classification at the end of the training | At the end of the sixth training week
  BRIEF-CORE SET OF THE ICF-CY (International Classification of Functioning, Disability and Health)
Change from baseline Functioning, Disability and Health classification at six months | At 6 months
  BRIEF-CORE SET OF THE ICF-CY (International Classification of Functioning, Disability and Health)
Change from baseline Functioning, Disability and Health classification at one year | At one year
  BRIEF-CORE SET OF THE ICF-CY (International Classification of Functioning, Disability and Health)

CONTACTS AND LOCATIONS:
Overall Officials: Jimena Quinzaños, MSc, Principal Investigator — Instituto Nacional de Rehabilitacion; Ivett Quiñones, PHD, Study Director — Instituto Nacional de Rehabilitacion
Locations (1):
- Instituto Nacional de Rehabilitación, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data could be available by e-mail and in order to ensure confidentiality they will be masked
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years from the beginning
Access Criteria: Authorization by e-mail

REFERENCES:
- [Background] Swinnen E, Duerinck S, Baeyens JP, Meeusen R, Kerckhofs E. Effectiveness of robot-assisted gait training in persons with spinal cord injury: a systematic review. J Rehabil Med. 2010 Jun;42(6):520-6. doi: 10.2340/16501977-0538. PMID 20549155
- [Background] Morawietz C, Moffat F. Effects of locomotor training after incomplete spinal cord injury: a systematic review. Arch Phys Med Rehabil. 2013 Nov;94(11):2297-308. doi: 10.1016/j.apmr.2013.06.023. Epub 2013 Jul 9. PMID 23850614
- [Background] Lucareli PR, Lima MO, Lima FP, de Almeida JG, Brech GC, D'Andrea Greve JM. Gait analysis following treadmill training with body weight support versus conventional physical therapy: a prospective randomized controlled single blind study. Spinal Cord. 2011 Sep;49(9):1001-7. doi: 10.1038/sc.2011.37. Epub 2011 May 3. PMID 21537338
- [Background] Colombo G, Wirz M, Dietz V. Driven gait orthosis for improvement of locomotor training in paraplegic patients. Spinal Cord. 2001 May;39(5):252-5. doi: 10.1038/sj.sc.3101154. PMID 11438840
- [Background] de Leon RD, Roy RR, Edgerton VR. Is the recovery of stepping following spinal cord injury mediated by modifying existing neural pathways or by generating new pathways? A perspective. Phys Ther. 2001 Dec;81(12):1904-11. PMID 11736625
- [Background] Threlkeld AJ, Cooper LD, Monger BP, Craven AN, Haupt HG. Temporospatial and kinematic gait alterations during treadmill walking with body weight suspension. Gait Posture. 2003 Jun;17(3):235-45. doi: 10.1016/s0966-6362(02)00105-4. PMID 12770637
- [Background] Dobkin B, Apple D, Barbeau H, Basso M, Behrman A, Deforge D, Ditunno J, Dudley G, Elashoff R, Fugate L, Harkema S, Saulino M, Scott M; Spinal Cord Injury Locomotor Trial Group. Weight-supported treadmill vs over-ground training for walking after acute incomplete SCI. Neurology. 2006 Feb 28;66(4):484-93. doi: 10.1212/01.wnl.0000202600.72018.39. PMID 16505299
- [Background] Scivoletto G, Tamburella F, Laurenza L, Torre M, Molinari M. Who is going to walk? A review of the factors influencing walking recovery after spinal cord injury. Front Hum Neurosci. 2014 Mar 13;8:141. doi: 10.3389/fnhum.2014.00141. eCollection 2014. PMID 24659962
- [Background] Manns PJ, Chad KE. Determining the relation between quality of life, handicap, fitness, and physical activity for persons with spinal cord injury. Arch Phys Med Rehabil. 1999 Dec;80(12):1566-71. doi: 10.1016/s0003-9993(99)90331-3. PMID 10597807
- [Background] Putzke JD, Richards JS, Hicken BL, DeVivo MJ. Predictors of life satisfaction: a spinal cord injury cohort study. Arch Phys Med Rehabil. 2002 Apr;83(4):555-61. doi: 10.1053/apmr.2002.31173. PMID 11932861
- [Background] Villiger M, Grabher P, Hepp-Reymond MC, Kiper D, Curt A, Bolliger M, Hotz-Boendermaker S, Kollias S, Eng K, Freund P. Relationship between structural brainstem and brain plasticity and lower-limb training in spinal cord injury: a longitudinal pilot study. Front Hum Neurosci. 2015 May 6;9:254. doi: 10.3389/fnhum.2015.00254. eCollection 2015. PMID 25999842
- [Result] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Result] Kirchberger I, Cieza A, Biering-Sorensen F, Baumberger M, Charlifue S, Post MW, Campbell R, Kovindha A, Ring H, Sinnott A, Kostanjsek N, Stucki G. ICF Core Sets for individuals with spinal cord injury in the early post-acute context. Spinal Cord. 2010 Apr;48(4):297-304. doi: 10.1038/sc.2009.128. Epub 2009 Sep 29. PMID 19786973
- [Result] Zarco-Perinan MJ, Barrera-Chacon MJ, Garcia-Obrero I, Mendez-Ferrer JB, Alarcon LE, Echevarria-Ruiz de Vargas C. Development of the Spanish version of the Spinal Cord Independence Measure version III: cross-cultural adaptation and reliability and validity study. Disabil Rehabil. 2014;36(19):1644-51. doi: 10.3109/09638288.2013.864713. Epub 2013 Dec 9. PMID 24320025
- [Result] Behrman AL, Lawless-Dixon AR, Davis SB, Bowden MG, Nair P, Phadke C, Hannold EM, Plummer P, Harkema SJ. Locomotor training progression and outcomes after incomplete spinal cord injury. Phys Ther. 2005 Dec;85(12):1356-71. PMID 16305274